CLINICAL TRIAL: NCT06896019
Title: The Association Mechanism Between the Microbiome and the Development of Community Pneumonia Was Studied Based on the Analysis of Pulmonary Microbiota - Host Interaction Network
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-628-01
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-08

CONDITIONS: Community Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAP
  Interventions: Diagnostic Test: Community Pneumonia

INTERVENTIONS:
Diagnostic Test: Community Pneumonia — The BALF of CAP patients

SUMMARY:
1. The difference of lung flora between the healthy group and the CAP group was compared, and the core flora involved in the development of CAP was identified.
2. To predict the metabolites associated with CAP.
3. Identification of genes related to immune response in CAP.
4. Construct the pulmonary microbiota - host interaction network with metabolites as the link.

ELIGIBILITY:
Inclusion Criteria:

* According to the CAP clinical diagnostic criteria in the Guidelines for the Diagnosis and Treatment of Community-Acquired Pneumonia in Adults in China (2016 edition), cases eligible for community-acquired pneumonia were included and screened.

Exclusion Criteria:

* Alveolar lavage fluid samples without electronic bronchoscopy were excluded for mNGS etiological examination of the case.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Community Pneumonia | 1 weeks
  mNGS

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sent Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No